CLINICAL TRIAL: NCT02255838
Title: Evaluation of a Disposable Flexible Bronchoscope, (aScope IV) a Randomized, Controlled, Cross-over Trial
Brief Title: Evaluation of a Disposable Flexible Bronchoscope, aScope IV
Acronym: EVAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment, outdated material
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rainer Lenhardt, MD, MBA, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 14.0689
Record Dates: First submitted 2014-09-24; First posted 2014-10-03 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Insufficiency; Pneumonia; Atelectasis
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: The disposable aScope IV bronchoscope will be compared to the re-usable bronchoscope
Masking Description: A blinded investigator will view the bronchoscopy video and evaluate. The blinded investigator will use the same criteria the investigator who did the procedure used (Un-blinded) for the evaluation. Video will not indicate which scope was used and only indicate if it is the right or left lung they are viewing. Research coordinator will keep separate a file indicating which scope was used.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disposable bronchoscope first (aScope IV), then Reusable bronchoscope (Storz 8402 2x) (Experimental): the bronchoscope will be re-inserted and advanced to the basal segmental bronchi of the right lower lobe. The tip of the bronchoscope will be brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml will be administered. The flow of saline will be observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction will be applied to collect the lavage specimen in the collection trap. This step will be repeated 4 more times (total of 80ml) to obtain an adequate specimen.
  Interventions: Device: Bronchoscope disposable (aScope 4)
- Reusable bronchoscope first (Storz 8402 2x), then Disposable bronchoscope (aScope IV) (Active Comparator): the bronchoscope will be re-inserted and advanced to the basal segmental bronchi of the right lower lobe. The tip of the bronchoscope will be brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml will be administered. The flow of saline will be observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction will be applied to collect the lavage specimen in the collection trap. This step will be repeated 4 more times (total of 80ml) to obtain an adequate specimen.
  Interventions: Device: Bronchoscope reusable (Storz 8402 2x)

INTERVENTIONS:
Device: Bronchoscope reusable (Storz 8402 2x) — Bronchoscopy and alveolar lavage
  Other Names: Storz 8402 2x (Storz, El Segundo, CA)
  Arms: Reusable bronchoscope first (Storz 8402 2x), then Disposable bronchoscope (aScope IV)
Device: Bronchoscope disposable (aScope 4) — Bronchoscopy and alveolar lavage
  Other Names: aScope 4 (Ambu, Glen Burnie, MD)
  Arms: Disposable bronchoscope first (aScope IV), then Reusable bronchoscope (Storz 8402 2x)

SUMMARY:
Flexible bronchoscopes are typically reusable and therefore need high level disinfection to prevent inadvertent spread of microbial pathogens from patient to patient. The process of disinfection is time consuming and expensive. Moreover, a bronchoscope being processed may not be readily available for another patient. One solution to this problem was to use a single use disposable sheath that covers a flexible bronchoscope protecting all surfaces of the bronchoscope.(Colt, Beamis, Harrell, & Mathur, 2000). Another way to eliminate potential hazards with a reusable bronchoscope is the use of a disposable bronchoscope. Such a disposable bronchoscope has been developed (Ambu aScope, Ambu, Glen Burnie, MD) and has been used successfully for intubations in manikins(Scutt et al., 2011) and patients. (Kristensen & Fredensborg, 2013; Pujol, López, & Valero, 2010; Tvede, Kristensen, & Nyhus-Andreasen, 2012). Further advancement in the imaging and handling of this disposable flexible bronchoscope now allows for the purpose of bronchoscopy and broncho-alveolar lavage in critically ill patients with pulmonary compromise. (FDA approval: 05-11-2013 date)

The aim of the study is to compare image clarity, suction capacity, and handling performance of a reusable flexible bronchoscope to the disposable flexible bronchoscope. In addition, the investigators intend to perform a cost analysis.

DETAILED DESCRIPTION:
Description

Patients will be monitored by standard NIBP or invasive arterial lines, ECG and oxygen saturation. All patients are intubated due to their respiratory insufficiency or for airway protection. Patients will be anesthetized for the procedure. Anesthesia will be induced with versed 2mg, fentanyl 100 µg and paralyzed with 0.1mg/kg vecuronium. Anesthesia will be maintained with propofol infusion 50-150 µg/kg/min.

Study Procedures All patients will be under general anesthesia. Standard monitoring will be applied. This includes a blood pressure cuff or an arterial line, EKG and a pulse-oximeter. Patients will receive 2 mg/kg propofol, 1µg/kg fentanyl and 0.1mg/kg vecuronium for the procedure. After induction of anesthesia the FiO2 will be turned to 1.0 and a bronchoscopy adaptor will be interposed in the breathing circuit next to the endotracheal tube. Patients will be randomized to receiving either the non-disposable bronchoscope (Storz 8402 2x, El Segundo, CA) or the single use aScope 3 first. After randomization, bronchoscopy will be started with an inspection of the trachea and carina. Next the right lung bronchial tree will be inspected systematically beginning with the right upper lobe, following with the right middle lobe and finishing with the right lower lobe. All segmental bronchi will be inspected and cleaned by suction as deemed necessary. The bronchoscope will then be removed from the bronchial tree and rinsed with saline Subsequently, the bronchoscope will be re-inserted and advanced to the basal segmental bronchi of the right lower lobe. The tip of the bronchoscope will be brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml will be administered. The flow of saline will be observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction will be applied to collect the lavage specimen in the collection trap. This step will be repeated 4 more times (total of 80ml) to obtain an adequate specimen. The same procedure will be repeated on the left lung using the alternate bronchoscope according to randomization. At the end of the procedure, a chest radiograph will be obtained to rule out pneumothorax.

Measurements

Before starting the procedure the set up time of each bronchoscope will be recorded. The view, image, and light of each bronchoscope will be assessed, then the inspection of the upper lobe segmental bronchi will be conducted. The time of lavage and suctioning until no more specimen can be collected will be measured. The volume of the obtained specimen will be measured. The specimen will be evaluated by a blinded observer after the procedure is completed.(clear fluids, mucous secretions, viscous secretions, pus, blood etc). The blinded observer will evaluate the quality and quanity of the sample for obtaining cultures.The blinded observer will be an attending or resident from the infectious disease department.

The overall ease of handling will be rated directly after the procedure by the investigator. All bronchoscopies will be taped and view-clarity, image and light-brightness will be assessed by a second blinded observer. This blinder observer can be another investigator not present during the procedure or an internist who was not present and is part of the study team.

All assessments will be performed using a VAS scale of 0 to 10 cm as shown below. The investigator will mark directly on the scale.

We will only enroll patients who were admitted to a critical care unit at the University of Louisville and who are intubated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult 18 years old and older
2. Capable of giving informed consent or have an acceptable surrogate capable of giving legally authorized consent on the subject's behalf.
3. Indication of a diagnostic and or therapeutic bronchoscopy as determined by the attending critical care physician
4. Being cared for in the critical care units at the U of L Hospital

Exclusion Criteria:

1) Patient is moribund and a bronchoscopy is very unlikely to reduce impending mortality or can avert death

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD MBA, Principal Investigator — University of Louisville School of Medicine Department of Anesthesiology and Perioperative Medicine
Locations (1):
- University of Louisville School of Medicine, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellomo R, Tai E, Parkin G. Fibreoptic bronchoscopy in the critically ill: a prospective study of its diagnostic and therapeutic value. Anaesth Intensive Care. 1992 Nov;20(4):464-9. doi: 10.1177/0310057X9202000412. PMID 1463174
- [Background] Colt HG, Beamis JJ, Harrell JH, Mathur PM. Novel flexible bronchoscope and single-use disposable-sheath endoscope system. A preliminary technology evaluation. Chest. 2000 Jul;118(1):183-7. doi: 10.1378/chest.118.1.183. PMID 10893377
- [Background] Estella A. [Analysis of 208 flexible bronchoscopies performed in an intensive care unit]. Med Intensiva. 2012 Aug-Sep;36(6):396-401. doi: 10.1016/j.medin.2011.11.005. Epub 2011 Dec 20. Spanish. PMID 22192316
- [Background] Facciolongo N, Patelli M, Gasparini S, Lazzari Agli L, Salio M, Simonassi C, Del Prato B, Zanoni P. Incidence of complications in bronchoscopy. Multicentre prospective study of 20,986 bronchoscopies. Monaldi Arch Chest Dis. 2009 Mar;71(1):8-14. doi: 10.4081/monaldi.2009.370. PMID 19522159
- [Background] Georgiades G, Myrianthefs P, Venetsanou K, Kythreoti A, Kyroudi A, Kittas C, Baltopoulos G. Temperature and serum proinflammatory cytokine changes in patients with NSCLC after BAL. Lung. 2003;181(1):35-47. doi: 10.1007/s00408-003-1001-6. PMID 12879338
- [Background] Huang YC, Bassett MA, Levin D, Montilla T, Ghio AJ. Acute phase reaction in healthy volunteers after bronchoscopy with lavage. Chest. 2006 Jun;129(6):1565-9. doi: 10.1378/chest.129.6.1565. PMID 16778276
- [Background] Ikeda S, Yanai N, Ishikawa S. Flexible bronchofiberscope. Keio J Med. 1968 Mar;17(1):1-16. doi: 10.2302/kjm.17.1. No abstract available. PMID 5674435
- [Background] Kreider ME, Lipson DA. Bronchoscopy for atelectasis in the ICU: a case report and review of the literature. Chest. 2003 Jul;124(1):344-50. doi: 10.1378/chest.124.1.344. PMID 12853543
- [Background] Kristensen MS, Fredensborg BB. The disposable Ambu aScope vs. a conventional flexible videoscope for awake intubation -- a randomised study. Acta Anaesthesiol Scand. 2013 Aug;57(7):888-95. doi: 10.1111/aas.12094. Epub 2013 Mar 15. PMID 23495767
- [Background] Lucena CM, Martinez-Olondris P, Badia JR, Xaubet A, Ferrer M, Torres A, Agusti C. [Fiberoptic bronchoscopy in a respiratory intensive care unit]. Med Intensiva. 2012 Aug-Sep;36(6):389-95. doi: 10.1016/j.medin.2011.11.004. Epub 2011 Dec 22. Spanish. PMID 22195599
- [Background] Perkins GD, Chatterjie S, McAuley DF, Gao F, Thickett DR. Role of nonbronchoscopic lavage for investigating alveolar inflammation and permeability in acute respiratory distress syndrome. Crit Care Med. 2006 Jan;34(1):57-64. doi: 10.1097/01.ccm.0000190197.69945.c5. PMID 16374157
- [Background] Pujol E, Lopez AM, Valero R. Use of the Ambu((R)) aScope in 10 patients with predicted difficult intubation. Anaesthesia. 2010 Oct;65(10):1037-40. doi: 10.1111/j.1365-2044.2010.06477.x. PMID 20707786
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. Summary of the British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults. Thorax. 2013 Aug;68(8):786-7. doi: 10.1136/thoraxjnl-2013-203629. PMID 23842821
- [Background] Scutt S, Clark N, Cook TM, Smith C, Christmas T, Coppel L, Crewdson K. Evaluation of a single-use intubating videoscope (Ambu aScope ) in three airway training manikins for oral intubation, nasal intubation and intubation via three supraglottic airway devices. Anaesthesia. 2011 Apr;66(4):293-9. doi: 10.1111/j.1365-2044.2011.06647.x. Epub 2011 Feb 24. PMID 21401543
- [Background] Sharif-Kashani B, Shahabi P, Behzadnia N, Mohammad-Taheri Z, Mansouri D, Masjedi MR, Zargari L, Salimi Negad L. Incidence of fever and bacteriemia following flexible fiberoptic bronchoscopy: a prospective study. Acta Med Iran. 2010 Nov-Dec;48(6):385-8. PMID 21287478
- [Background] Steinberg KP, Mitchell DR, Maunder RJ, Milberg JA, Whitcomb ME, Hudson LD. Safety of bronchoalveolar lavage in patients with adult respiratory distress syndrome. Am Rev Respir Dis. 1993 Sep;148(3):556-61. doi: 10.1164/ajrccm/148.3.556. PMID 8368623
- [Background] Tsao TC, Tsai YH, Lan RS, Shieh WB, Lee CH. Treatment for collapsed lung in critically ill patients. Selective intrabronchial air insufflation using the fiberoptic bronchoscope. Chest. 1990 Feb;97(2):435-8. doi: 10.1378/chest.97.2.435. PMID 2298070
- [Background] Tvede MF, Kristensen MS, Nyhus-Andreasen M. A cost analysis of reusable and disposable flexible optical scopes for intubation. Acta Anaesthesiol Scand. 2012 May;56(5):577-84. doi: 10.1111/j.1399-6576.2012.02653.x. Epub 2012 Feb 16. PMID 22338623
- [Background] Um SW, Choi CM, Lee CT, Kim YW, Han SK, Shim YS, Yoo CG. Prospective analysis of clinical characteristics and risk factors of postbronchoscopy fever. Chest. 2004 Mar;125(3):945-52. doi: 10.1378/chest.125.3.945. PMID 15006953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: period August 8, 2015 to July 8, 2017 location: ICU
Groups:
- Disposable Bronchoscope First (aScope IV), Then Reusable Bronchoscope (Storz 8402 2x): Randomly controlled, either the disposable bronchoscope (aScope 4) was inserted first into the trachea and advanced into the right lung. Subsequently, a reusable bronchoscope (Storz 8402) was inserted into the trachea and advanced into the left lung. If randomization assigned the reusable bronchoscope to be inserted first, then the reusable bronchoscope was inserted into the trachea and advanced into the right lung first followed by insertion of the disposable bronchoscope and advancement into the left lung. The subsequent procedure was identical for both parts of this crossover trial and is described as follows: After insertion of the bronchoscope into the bronchial tree the scope was advanced to the basal segmental bronchi of the right or left lower lobe. The tip of the bronchoscope was brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml was administered. The flow of saline was observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction was applied to collect the lavage specimen in the collection trap. This step was repeated 4 more times (total of 80 ml) to obtain an adequate specimen.
- Reusable Bronchoscope First (Storz 8402 2x), Then Disposable Bronchoscope (aScope IV): Randomly controlled, either the reusable bronchoscope (Storz 8402) was inserted first into the trachea and advanced into the right lung. Subsequently, disposable bronchoscope (aScope 4) was inserted into the trachea and advanced into the left lung. If randomization assigned the reusable bronchoscope to be inserted first, then the reusable bronchoscope was inserted into the trachea and advanced into the right lung first followed by insertion of the disposable bronchoscope and advancement into the left lung. The subsequent procedure was identical for both parts of this crossover trial and is described as follows: After insertion of the bronchoscope into the bronchial tree the scope was advanced to the basal segmental bronchi of the right or left lower lobe. The tip of the bronchoscope was brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml was administered. The flow of saline was observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction was applied to collect the lavage specimen in the collection trap. This step was repeated 4 more times (total of 80 ml) to obtain an adequate specimen.
Period: Overall Study
Arm/Group | Disposable Bronchoscope First (aScope IV), Then Reusable Bronchoscope (Storz 8402 2x) | Reusable Bronchoscope First (Storz 8402 2x), Then Disposable Bronchoscope (aScope IV)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants were randomized to receive both intervention in a sequential order, per a cross-over study design
Groups:
- Disposable Bronchoscope Insertion Followed by Reusable Bronchoscope Insertion or Vice Versa: Randomly controlled, either the disposable bronchoscope (aScope 4) was inserted first into the trachea and advanced into the right lung. Subsequently, a reusable bronchoscope (Storz 8402) was inserted into the trachea and advanced into the left lung. If randomization assigned the reusable bronchoscope to be inserted first, then the reusable bronchoscope was inserted into the trachea and advanced into the right lung first followed by insertion of the disposable bronchoscope and advancement into the left lung. The subsequent procedure was identical for both parts of this crossover trial and is described as follows: After insertion of the bronchoscope into the bronchial tree the scope was advanced to the basal segmental bronchi of the right or left lower lobe. The tip of the bronchoscope was brought into wedge position in one of the basal segments for broncho-alveolar lavage (BAL). A saline flush of 20 ml was administered. The flow of saline was observed at the distal tip of the bronchoscope. After 10 seconds of maintaining a wedge position, gentle suction was applied to collect the lavage specimen in the collection trap. This step was repeated 4 more times (total of 80 ml) to obtain an adequate specimen.
Arm/Group | Disposable Bronchoscope Insertion Followed by Reusable Bronchoscope Insertion or Vice Versa
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Visualization of Two Different Flexible Bronchoscopes; a Disposable and a Reusable Bronchoscope
Description: Visualization of the two bronchoscopes was measured by using a qualitative scale from 0 to 10; 0 being classified as "cannot be evaluated" and 10 being assessed as optimal visualization
Time Frame: 10 to 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Bronchoscope Disposable, aScope IV: Randomly controlled, the disposable bronchoscope (aScope 4) was inserted into the trachea and advanced into the right lung or the disposable bronchoscope was inserted as the second bronchoscope into the left lung.
- Reusable Bronchoscope (Storz 8402): Randomly controlled, the reusable bronchoscope (Storz 8402) was inserted into the trachea and advanced into the right lung or the reusable bronchoscope was inserted as the second bronchoscope into the left lung.
Arm/Group | Bronchoscope Disposable, aScope IV | Reusable Bronchoscope (Storz 8402)
Number analyzed (Participants) | 12 | 12
score on a scale | 7.5 (1.2) | 8.0 (0.7)
Statistical Analysis 1: Comparison: Bronchoscope Disposable, aScope IV vs Reusable Bronchoscope (Storz 8402); Test type: Superiority; p < 0.05, t-test, 2 sided; paired t-test

2. Primary Outcome: Evaluation of the Handling of Two Different Flexible Bronchoscopes, a Disposable and a Reusable Bronchoscope
Description: Handling of the two bronchoscopes using a qualitative scale from 0 to 10; 0 being classified as "cannot be evaluated" and 10 being assessed as optimal visualization
Time Frame: 10-30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Reusable Bronchoscope(Storz 8402): Randomly controlled, the reusable bronchoscope (Storz 8402) was inserted into the trachea and advanced into the right lung or the reusable bronchoscope was inserted as the second bronchoscope into the left lung.
Arm/Group | Bronchoscope Disposable, aScope IV | Reusable Bronchoscope(Storz 8402)
Number analyzed (Participants) | 12 | 12
score on a scale | 8.0 (1.5) | 8.0 (1.1)

3. Secondary Outcome: Evaluation of Ability to Suction With Two Different Flexible Bronchoscopes, a Disposable and a Reusable Bronchoscope
Description: Measured suction capability by volume retrieved after broncho-alveolar lavage with 10 ml of saline, measured in ml
Time Frame: 10-30 minutes
Measure: Mean (Standard Deviation); unit: milliliter
Groups:
- Bronchoscope Reusable Storz 8402 2x: Randomly controlled, the reusable bronchoscope (Storz 8402) was inserted into the trachea and advanced into the right lung or the reusable bronchoscope was inserted as the second bronchoscope into the left lung.
Arm/Group | Bronchoscope Disposable, aScope IV | Bronchoscope Reusable Storz 8402 2x
Number analyzed (Participants) | 12 | 12
milliliter | 5.4 (0.9) | 5.3 (1.0)

4. Secondary Outcome: Evaluation of Flexibility of Two Different Flexible Bronchoscopes, a Disposable and a Reusable Bronchoscope
Description: Flexibility of the two bronchoscopes was measured by using a qualitative scale from 0 to 10; 0 being classified as "cannot be evaluated" and 10 being assessed as optimal flexibility
Time Frame: 10-30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bronchoscope Disposable, aScope IV | Bronchoscope Reusable Storz 8402 2x
Number analyzed (Participants) | 12 | 12
score on a scale | 8.7 (10) | 7.4 (1.3)

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: routine bronchoscopies in the ICU, potential adverse events were observed during the study period of 10-30 minutes and for one hour after the bronchoscopy
Groups:
- Disposable Bronchoscope First (aScope IV), Then Reusable Bronchoscope (Storz 8402 2x); Reusable Bronchoscope First (Storz 8402 2x), Then Disposable Bronchoscope (aScope IV): no adverse events
Arm/Group | Disposable Bronchoscope First (aScope IV), Then Reusable Bronchoscope (Storz 8402 2x) | Reusable Bronchoscope First (Storz 8402 2x), Then Disposable Bronchoscope (aScope IV)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-06-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT02255838/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02255838/ICF_001.pdf